CLINICAL TRIAL: NCT06295146
Title: Improving Manual Wheelchair Skills Through Remote Training
Brief Title: Virtual Peer Coaching in Manual Wheelchair Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lynn Worobey, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY23050075
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Wheelchair; Paraplegia; Spinal Cord Injury; Tetraplegia/Tetraparesis; Spinal Cord Injuries (SCI)
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Intervention Model Description: For trainees, we will use a randomized, single-blinded, two-period cross-over study design for Groups 1 and 2. Participants will complete baseline assessments and then be randomized to either Group 1 or Group 2. After we have completed enrollment for Groups 1 and 2 (N=40 per group) we will enroll participants into Group 3 ( N=40 per group).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active intervention (intervention A) (Experimental): Active intervention (intervention A) which will include training through peer coaching
  Interventions: Other: Intervention A: 1-on-1 wheelchair skills training by a peer coach
- Waitlist control group (Active Comparator): Waitlist control group that will receive the same intervention A but at 6 months
  Interventions: Other: Intervention A: 1-on-1 wheelchair skills training by a peer coach
- Self-study intervention (Active Comparator): Self-study intervention with review of educational materials
  Interventions: Other: Intervention B: Training via educational videos

INTERVENTIONS:
Other: Intervention A: 1-on-1 wheelchair skills training by a peer coach — Trainees will engage in 1:1 virtual zoom meetings facilitated by the study team scheduled weekly for 6 sessions with the opportunity for 2 makeup sessions. Sessions will last approximately 30 minutes and may include goal setting, review of progress, instruction, and "homework" of prescribed content for trainees to review. Participants may upload videos of themselves completing skills through Qualtrics to get feedback.
  Arms: Active intervention (intervention A); Waitlist control group
Other: Intervention B: Training via educational videos — Intervention B will be a series of educational videos that participants review and then are encouraged to the practice the skills. Participants will have access to the materials for 8 weeks. Group 3 will have access to approximately 3 hours of wheelchair skills video training content. Actual viewing time will depend upon the individual's training goal. While they will receive a weekly reminder about practicing, there is no prescribed frequency for how often they should be practicing the skills in the videos.
  Arms: Self-study intervention

SUMMARY:
The objective of this study is to determine the effectiveness of remote manual wheelchair skills training program. First, peer coaches will be enrolled and trained. Then, trainees will be enrolled into one of three interventions: intervention with remote feedback (Group 1), wait list control group (Group 2), and structured self-study (Group 3).

DETAILED DESCRIPTION:
For peer coaches:

Coaches will complete the following measures pre and post training:

* Demographic questionnaire
* Self-Efficacy on Assessing, Training, and Spotting (SEATS)
* Feedback survey

Prior to coaching trainees, coaches will undergo three training programs as follows:

* Virtual training through zoom on peer mentoring
* Research ethics training
* Wheelchair skills training

It will be verified that peer coaches possess the needed skills by administering the SEATS following training. A score of 5 (completely confident) for each training item will be required to advance to the peer coaching sessions.

For peer coaching, coaches will lead six 1:1 virtual zoom meetings with each trainee they are matched with. Sessions may include goal setting, review of progress, instruction, and "homework" of prescribed content for trainees to review. For each training session coaches will complete a session log.

For trainees:

Baseline questionnaires will include:

* Demographic questionnaire
* Wheelchair setup questionnaire
* Wheelchair Skills Test Questionnaire (WST-Q)
* Goal Attainment Scale (GAS) (Group 1,3 only)
* Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF) Mobility
* Wheelchair Outcome Measure (WhOM) Satisfaction with Participation in Meaningful Activities
* Life Space Assessment (LSA)
* Online Learning Readiness Scale (OLRS)
* Moorong Self-Efficacy Scale (MSES)
* Referral Source
* Wheelchair Skills Training Questionnaire
* Wheelchair skills training outside of study

Group Specific Activities

Groups 1 and 2 will complete intervention A following baseline and 6-month assessments, respectively. Group 3 will complete intervention B. Participants in all groups will select what goals are important to them. They are not required to complete training in all skills, only to have at least 5 skills with relevant training goals.

Intervention A Trainees will engage in 1:1 virtual zoom meetings facilitated by the study team scheduled weekly for 6 sessions with the opportunity for 2 makeup sessions. Sessions may include goal setting, review of progress, instruction, and "homework" of prescribed content for trainees to review. Participants may upload videos of themselves completing skills through Qualtrics to get feedback.

Skills targeted by the intervention -

1. opening/closing doors
2. picking up an object from the ground
3. getting over a gap
4. getting over a threshold
5. up a low curb
6. down a low curb
7. up a high curb
8. down a high curb
9. performing a stationary wheelie
10. up a steep incline
11. down a steep incline
12. getting up stairs
13. getting down stairs
14. uneven transfers
15. floor-to-chair transfer
16. folding and unfolding wheelchair

Intervention B Intervention B will be a series of educational videos that participants review and then are encouraged to practice the skills. Participants will have access to the materials for 8 weeks. Group 3 will have access to approximately 3 hours of wheelchair skills video training content. Actual viewing time will depend upon the individual's training goal. While they will receive a weekly reminder about practicing, there is no prescribed frequency for how often they should be practicing the skills in the videos.

All participants will complete 2-month follow-up. This will include the following questionnaires:

Baseline questionnaires will include:

* Wheelchair setup questionnaire
* Wheelchair skills training outside of study survey
* Wheelchair Skills Test Questionnaire (WST-Q)
* Goal Attainment Scale (GAS) - groups 1 and 3 only
* Feedback Survey - groups 1 and 3 only
* Wheelchair skills training outside of study

All participants will complete 6-month follow-up. This will include the following questionnaires:

* Wheelchair setup questionnaire
* Wheelchair skills training outside of study survey
* Wheelchair Skills Test Questionnaire (WST-Q)
* Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF) Mobility
* Wheelchair Outcome Measure (WhOM) Satisfaction with Participation in Meaningful Activities
* Life Space Assessment (LSA)
* Wheelchair skills training outside of study

Groups 2 will then cross-over to complete intervention A.

All participants will complete 8-month follow-up. This will include the following questionnaires:

* Wheelchair setup questionnaire
* Wheelchair skills training outside of study survey
* Wheelchair Skills Test Questionnaire (WST-Q)
* Goal Attainment Scale (GAS) - group 2 only
* Feedback Survey - group 2 only
* Wheelchair skills training outside of study

All participants will complete 12-month follow-up. This will include the following questionnaires:

* Wheelchair setup questionnaire
* Wheelchair Skills Test Questionnaire (WST-Q)
* Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF) Mobility
* Wheelchair Outcome Measure (WhOM) Satisfaction with Participation in Meaningful Activities
* Life Space Assessment (LSA)
* Wheelchair skills training outside of study

Follow-up windows will be within approximately 2 weeks before/after the follow-up date. Participants will be asked to select two preferred methods of contact for follow-up reminders that will be sent between timepoints.

Spotters are required for trainee participation in the study. Prior to the start of the study, spotters will be required to watch a series of training videos about safe spotting.

ELIGIBILITY:
Inclusion Criteria:

Coaches:

* At least 18 years old
* Non-progressive SCI
* Able to speak and read English
* Reside in the community
* Independently use a manual wheelchair for at least 50% of mobility

Coaches with paraplegia:

- Able to complete all skills targeted by the intervention, except stair ascent, (WST-Q item scores 2) independently.

Coaches with tetraplegia:

- Able to complete all skills targeted by the intervention with or without assistance

Trainees:

* At least 18 years old
* Non-progressive SCI
* Able to speak and read English
* Reside in the community
* Independently use a manual wheelchair for 50% of mobility
* Access to an Internet-ready device with video capabilities.
* Access to a spotter for practicing wheelchair skills
* Desire training for at least 5 of the 16 skills targeted by the training program

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Capacity, confidence, and performance of wheelchair skills will improve following training | 6 months
  Compare the results of the Wheelchair Skills Test Questionnaire (WST-Q) between groups.
  The WST-Q is a self report measure of capacity (ability to complete), confidence, and performance (frequency of completing) wheelchair skills. The WST-Q will measured for each of 16 skills targeted in the training and a total score for each domain will be calculated.

SECONDARY OUTCOMES:
Wheelchair Skills Test Questionnaire (WST-Q) improvement from baseline following training | Post-training (2 mo assessment for groups 1 and 3; 8 mo assessment for group 2)
  Compare the results of the WST-Q taken after training to the beginning of study.
Wheelchair Skills Test Questionnaire (WST-Q) improvement from baseline (6 months) | 6 months post training (6 mo assessment for groups 1 and 3; 12 mo assessment for group 2)
  Compare the results of the WST-Q taken 6 months after training to the beginning of study.
Wheelchair Skills Test Questionnaire (WST-Q) improvement from baseline (12 months) | 1 year
  Compare the results of the WST-Q taken 12 months after the beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
Goal Attainment Scale (GAS) improvement from baseline (post training) | Post-training (2 mo assessment for groups 1 and 3; 8 mo assessment for group 2)
  Compare the results of the GAS taken post training to results at beginning of study.
  For GAS, the wheelchair trainer and trainee will set specific, measurable, attainable, realistic, and time related individual goals. The goals are weighted for importance (0=not at all important, to 3=very important) and difficulty (0=not at all difficult, to 3=very difficult). The wheelchair skill is performed and rated. Possible performance level scores: +2 (much more than expected), +1 (more than expected), 0 expected level, -1 (less than expected), or -2 (much less than expected).
Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF) Mobility improvement (6 months) | 6 months
  Compare the results of the CHART taken at 6 months to results at beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
  The CHART is designed as an interview tool, which can be administered face-to-face or by telephone. CHART produces an index of handicap. It is possible to score more than 100 on most of the subscales, however a maximum of 100 points has been allowed, indicating no handicap in that dimension. Scoring takes into account: physical independence, cognitive independence, mobility, occupation, social integration, and economic self-sufficiency.
Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF) Mobility improvement (1 year) | 1 year
  Compare the results of the CHART taken at 1 year to results at beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
Wheelchair Outcome Measure (WhOM) Satisfaction with Participation in Meaningful Activities after baseline (6 months) | 6 months
  Compare the results of the WhOM taken at 6 months to results at beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
  The WhOM is a client-centred measure of wheelchair and seating system intervention.The WhOM is a two part questionnaire which can be administered by a therapist in under 30 minutes, focused on participation outcomes as identified by the participants.
  Participants identify their participation outcome goals (i.e. specific things that they want to do and achieve) at home and in the community, and they then rate the importance (Imp) of the goals and satisfaction (Sat) with their performance in reaching their goals. Imp and Sat are rated (0-10) for each identified activity. Sat x Imp score (0-100) for each activity is the product of the two values. Mean Sat and mean Sat x Imp scores are the means of the respective activity scores.
Wheelchair Outcome Measure (WhOM) Satisfaction with Participation in Meaningful Activities after baseline (1 year) | 1 year
  Compare the results of the WhOM taken at 1 year to results at beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
Life Space Assessment (LSA) improvement from baseline (6 months) | 6 months
  Compare the results of the LSA taken at 6 months to results at beginning of study. Group 1 will have received peer coaching, group 2 is the control group, and group 3 will have completed self-study using videos.
  The overall score for each life-space level and the total score are calculated by summing the scores. The total score ranges from 0 ("totally bed-bound") to 120 ("traveling out of town every day without assistance"). The LSA is positively scored, with higher scores indicating a larger life space.
Life Space Assessment (LSA) improvement from baseline (1 year) | 1 year
  Compare the results of the LSA taken at 1 year to results at beginning of study. Group 1 will have received peer coaching 6 months prior, group 2 will have received peer coaching most recently, and group 3 will have completed self-study using videos.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Worobey, PhD/DPT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States